CLINICAL TRIAL: NCT00217035
Title: Glutamine Enriched Total Parenteral Feeding and Proline Metabolism in Severely Burned Patients.
Status: Withdrawn | Type: Observational
Why Stopped: State of Mass. tightened regulations for making intravenous solutions for research subjects. Study was withdrawn and no participants were enrolled.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Ronald G. Tompkins, MD, ScD, Chief, Burn Service, Massachusetts General Hospital
Organization: National Institute of General Medical Sciences (NIGMS) (NIH)
Other Study IDs: 1999-P-008462; 2P50GM021700-27 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Burns
Keywords: parenteral nutrition; burn injury; stable isotopes; Proline Metabolic Kinetics; Ornithine Metabolic Kinetics; Glutamate Metabolic Kinetics; Glutamine Metabolic Kinetics
MeSH Terms: conditions — Burns; Hyperphagia | interventions — Glutamine; Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: TPN or TPN enriched with glutamine — Each patient undergoes two nutritional support periods either with or without Glutamine supplementation.
  Other Names: Nutritional Support; Amino Acid Composition

SUMMARY:
Proline is a non-essential amino acid that helps with collagen formation. Collagen is one of the main ingredients of skin, bone, tendons, and connective tissue. It is thought that proline becomes depleted in burn patients because it is being used in greater than normal quantities to help the injured skin and connective tissue heal. If this is true, then the body must look for alternate energy sources as proline becomes depleted.

This study aims to evaluate 1)the metabolic kinetics of the amino acids proline, glutamate, and ornithine and 2) the effects of glutamine supplemented total parenteral nutrition (TPN) on the metabolism of these amino acids.

DETAILED DESCRIPTION:
Proline is a nutritionally dispensable (non-essential) amino acid. Its synthesis and catabolism is via the pathway of ornithine and glutamate. The latter two amino acids serve as immediate precursors for proline, as well as metabolites. Ornithine is one of the intermediates for urea cycle. Glutamate is metabolically connected to tricarboxylic acid (TCA) cycle, the major cycle for energy production.

It is hypothesized that the significantly increased rates of net nitrogen loss and energy "production", as the consequence of the accelerated activities of both the urea and TCA cycles in burn injury "drain" both ornithine and glutamate, thus depleting tissues of the availability of proline. Hence, the de novo synthesis of proline is likely to be affected by the reduced availability of its major precursors: glutamate and ornithine. We further propose that increased supply of glutamine would increase the de novo synthesis of proline and / or spare the loss of proline via its metabolite glutamate. Hence, glutamine will be beneficial to the overall nutritional status of the burn patients.

ELIGIBILITY:
Inclusion Criteria:

Burn patients being treated at MGH Burn Unit with one or more of the following criteria: 1) >=5% TBSA; 2) inhalation injury; or 3) resting energy expenditure (REE) of >15% of the predicted Basal Metabolic Rate using the Harris-Benedict equation.

Must be receiving total parenteral nutrition in the course of their treatment.

Exclusion Criteria:

Patients with thyroid disease. Patients who are not hemodynamically stable or show unstable vital signs Patients at the stage of major organ failure, e.g. renal and/or liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1997-08; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
This is a study for measuring the protein kinetics for metabolism of the amino acids proline, glutamate, and ornithine. Kinetics will be derived from measurements on blood and air samples taken as part of the study. | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Tompkins, MD, ScD, Principal Investigator — MGH, Shriners Burn Hospital - Boston
Locations (1):
- Massachusetts General Hospital Burn Unit, Boston, Massachusetts, United States

REFERENCES:
- [Background] Tharakan JF, Yu YM, Zurakowski D, Roth RM, Young VR, Castillo L. Adaptation to a long term (4 weeks) arginine- and precursor (glutamate, proline and aspartate)-free diet. Clin Nutr. 2008 Aug;27(4):513-22. doi: 10.1016/j.clnu.2008.04.014. Epub 2008 Jun 30. PMID 18590940
- [Background] Yu YM, Ryan CM, Castillo L, Lu XM, Beaumier L, Tompkins RG, Young VR. Arginine and ornithine kinetics in severely burned patients: increased rate of arginine disposal. Am J Physiol Endocrinol Metab. 2001 Mar;280(3):E509-17. doi: 10.1152/ajpendo.2001.280.3.E509. PMID 11171607
- [Background] Castillo L, Ajami A, Branch S, Chapman TE, Yu YM, Burke JF, Young VR. Plasma arginine kinetics in adult man: response to an arginine-free diet. Metabolism. 1994 Jan;43(1):114-22. doi: 10.1016/0026-0495(94)90166-x. PMID 8289668
- [Background] Jaksic T, Wagner DA, Burke JF, Young VR. Proline metabolism in adult male burned patients and healthy control subjects. Am J Clin Nutr. 1991 Aug;54(2):408-13. doi: 10.1093/ajcn/54.2.408. PMID 1858705
- [Background] Jaksic T, Wagner DA, Burke JF, Young VR. Plasma proline kinetics and the regulation of proline synthesis in man. Metabolism. 1987 Nov;36(11):1040-6. doi: 10.1016/0026-0495(87)90023-0. PMID 3670073